CLINICAL TRIAL: NCT02965508
Title: Home-based Primary Care for Homebound Seniors: a Randomized Controlled Trial
Brief Title: Home-based Primary Care for Homebound Seniors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Data Safety Monitoring Board determined that the serious adverse event rate was higher among patients awaiting enrollment in the home-based primary care intervention compared to those who had initiated home-based primary care.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); NYU Langone Health (Other); University of California, San Francisco (Other); Visiting Nurse Service of New York (Other); The New Jewish Home (Unknown)
Responsible Party: Principal Investigator, Alex D Federman, Professor, Geriatrics and Palliative Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 15-0950; R01AG052557 (NIH)
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Home-bound Adults
Keywords: Home-bound; home-based primary care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Primary Care Arm (Experimental): Participants in this arm will be assigned a Mount Sinai Visiting Doctors primary care physician who makes a home based primary care visit.
  Interventions: Other: Home-based Primary Care
- Usual Care Arm (Active Comparator): Participants in this arm will receive the usual care at office based visits
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Home-based Primary Care — Care in the programs is inter-professional and team-based. Each physician leads a team charged with the care of a panel of patients and directs the team's activities. New patients are assigned a Mount Sinai Visiting Doctors (MSVD) primary care physician or the Chelsea Village House Calls Program (CVHCP) who makes an initial visit within 2 weeks of the patient's enrollment in the program. The primary care physician completes a comprehensive medical history and physical exam during the initial visit including standardized assessments of physical functioning and cognition. The primary care physician then provides ongoing management of the patients' acute and chronic health problems, including palliative and home hospice care when needed, every 2 to 12 weeks as determined on a case-by-case basis.
  Arms: Home-based Primary Care Arm
Other: Usual Care — Office based care
  Arms: Usual Care Arm

SUMMARY:
The objective of this pragmatic randomized controlled trial is to compare the impact of physician directed home-based primary care with office-based primary care on hospitalizations, symptom control, caregiver burden, healthcare costs and other outcomes for older homebound adults and to conduct a dissemination and implementation evaluation to support future home-based primary care adoption

DETAILED DESCRIPTION:
The objective of this study is to evaluate the impact of home-based primary care on outcomes for home-bound older adults, including hospitalization and emergency department (ED) visits, quality of life and symptom control, costs of care, and burden of care for their informal caregivers. A mixed methods dissemination and implementation evaluation of home-based primary care will also be conducted.

Over one million seniors in the U.S. have functional limitations that prevent them from receiving office-based primary care. As a result, home-bound adults typically experience poor disease control, high rates of hospitalization, and large healthcare expenditures resulting for hospitalizations and emergency department use. Few modes of healthcare delivery designed specifically for the home-bound have been studied, but observational data suggest that home-based primary care could improve outcomes and reduce spending for these highly vulnerable patients.

The investigators propose a pragmatic randomized controlled trial of home-based primary care vs. office-based primary care for home-bound older adults, with 3 Specific Aims: to compare the impact of home-based primary care and office-based primary care 1) on hospitalization and emergency department visit rates, symptom control and quality of life, and satisfaction with care among home-bound elders; 2) on care-giving burden among informal caregivers (e.g., family and friends); and 3) on healthcare expenditures for the home-bound. The hypothesis is that patients in home-based primary care and their caregivers will have better outcomes compared to office-based primary care patients.

The study embraces the concepts of a pragmatic trial design to facilitate the translation of study findings for practical clinical, systems, and health policy applications. The study team includes experts in aging related health services research, health economics, health policy, randomized clinical trials, and the medical and nursing care of home-bound older adults.

The proposed study would be the largest prospective study of home-bound older adults and the only randomized trial of home-based primary car for the home-bound. It would fill important knowledge gaps in our understanding of the effects of home-based primary care for the home-bound. The study is consistent with the Institute of Medicine's call for expanded research on comprehensive models of chronic care, including the multidisciplinary management of chronic diseases and the medical home concept.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years with Medicare
* Able to provide informed consent (patient or proxy)
* Permanently requires assistance in ≥2 activities of daily living
* Patient or proxy reports that patient is home-bound (leaves the home infrequently for non-medical purposes or cannot leave the home without assistance)
* ≥1 hospitalization in past 12 months
* Speaks English or Spanish
* Willingness to accept a home-based primary care physician as their primary care physician.

Exclusion Criteria:

* Patients must live in Manhattan, have access to a telephone 24 hours a day, 7 days a week, not be on hemodialysis, agree to open the door and allow access to the members of the team
* If there is any active drug use/sale or firearms in home, we exclude for safety reasons
* A 2-week prognosis will be based on the opinion of the patient's primary care provider or by consensus among physicians on the research team
* Patients in hospice at baseline
* Standard MSVD and CVHCP exclusion criteria also apply :(1) Patients must live in Manhattan, have access to a telephone 24/7, not be on hemodialysis, agree to open the door and allow access to the members of the team; (2) If there is any active drug use/sale or firearms in home, will exclude for safety reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Hospitalization | at 12 months
Incidence of ED visits | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex Federman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No